CLINICAL TRIAL: NCT06990932
Title: High Intensity Laser vs Instrument-assisted Soft Tissue Mobilization on Trapezius Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Adel Ahmed Abdelmoaty AboHashish, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ahmed-005701
Record Dates: First submitted 2025-05-18; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: High Intensity Laser; Instrument Assisted Soft Tissue Mobilization; Trapezius Muscle Strain; Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Intensity Laser (Experimental): this group consists of 20 subjects will receive conventional treatment combined with High-intensity laser therapy, three times per week for one month
  Interventions: Device: High Intensity Laser; Other: Conventional treatment
- Instrument-assisted soft tissue mobilization (Active Comparator): this group consists of 20 subjects will receive conventional treatment combined with Instrument-assisted soft tissue mobilization, three times per week for one month
  Interventions: Other: Instrument-assisted Soft Tissue Mobilization; Other: Conventional treatment
- conventional treatment (Active Comparator): this group consists of 20 subjects will receive conventional treatment only, three times per week for one month
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Device: High Intensity Laser — The therapeutic dose of laser therapy depends on power density, tissue color, and type. Darker skin may absorb the laser in the epidermal layer, but HILT can pass through without absorption. Research has improved power density and dose, with the World Association of Laser Therapy recommending a 5-7 J/cm2 dose for optimal therapeutic outcomes.
  Arms: High Intensity Laser
Other: Instrument-assisted Soft Tissue Mobilization — Instrument-assisted soft tissue mobilization is a popular alternative to traditional manual therapy techniques, derived from Cyriax cross-friction massage. It uses hard tools to manipulate soft tissue, varying in direction, force, and pattern, and allowing pressure to disperse to underlying tissues. Modern Instrument-assisted soft tissue mobilization instruments vary in material and design, and are used to improve musculoskeletal conditions and outcomes. Patients receive Instrument-assisted soft tissue mobilization with an M2T blade, positioned at a 45° angle, and instructed to apply an ice pack if experiencing burning sensations.
  Arms: Instrument-assisted soft tissue mobilization
Other: Conventional treatment — conventional physical therapy, which includes ultrasound, isometric neck exercises, chin tucks, stretching of neck muscles, and neck stabilization exercises, were used for groups A, B and C

SUMMARY:
The purpose of the study was to

1. Investigate the effect of high-intensity laser therapy versus Instrument-assisted soft tissue mobilization on pain level in patients with myofascial pain syndrome of upper trapezius muscle.
2. Investigate the effect of High intensity laser therapy versus Instrument-assisted soft tissue mobilization on ROM in patients with myofascial pain syndrome of upper trapezius muscle

DETAILED DESCRIPTION:
Myofascial pain syndrome is a common musculoskeletal pain affecting 30% of patients in primary care. It is characterized by trigger points in the upper trapezius muscle, which is linked to neck and shoulder pain. Non-invasive treatments like exercises, manipulation, and physical agents have been suggested for managing neck pain. Laser therapy, including low-level and high-intensity, has been found effective in reducing pain intensity and improving functional activity. Instrument-assisted soft tissue mobilization is another technique used to treat Myofascial pain syndrome. Instrument-assisted soft tissue mobilization stimulates connective tissue remodeling, resorbing excessive fibrosis, and promoting collagen repair and regeneration. The study aims to investigate the effect of high intensity laser therapy versus Instrument-assisted soft tissue mobilization in treating Myofascial pain syndrome of the upper trapezius muscle.

ELIGIBILITY:
Inclusion Criteria:

1. The patient age ranged from 20 to 50 years
2. Presence of myofascial trigger points in the upper trapezius muscle
3. Having neck discomfort symptoms that were triggered by certain neck positions and by palpating the cervical musculature for at least three months
4. Patient willing and able to participate in an exercise program safely

Exclusion Criteria:

1. medical red flag history (such as tumour, fracture, metabolic diseases, rheumatoid arthritis and osteoporosis)
2. Neck pain with cervical radiculopathy or neck pain associated with externalized cervical disc herniation.
3. If the patient had previous surgery in the neck area (irrespective of the reason for the operation)
4. Neck pain accompanied by vertigo caused by vertebra basilar insufficiency or accompanied by non-cervicogenic headaches

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Assessment of change of pain intensity | At baseline and after 1 month
  The Visual Analog Scale is a self-reported pain measurement scale with a 10-cm line labeling extreme pain levels. It is valid, reliable, and suitable for clinical practice, especially for individuals over 18. Studies have shown moderate to strong correlations for VAS validity in pain measurement.

SECONDARY OUTCOMES:
Assessment of change of pressure pain threshold | At baseline and after 1 month
  A pressure algometer is a reliable tool for determining local pressure pain threshold (PPT) in different pain syndromes. It is a force gauge calibrated in kg/cm2 and has a range of 0-10 kg/cm2. A manual pressure algometer will be used to measure pain threshold for upper trapezius fibers, with repeated measurements to improve reliability.
Assessment of change of Cervical range of motion | At baseline and after 1 month
  The CROM device is a lightweight, comfortable, and secure device that adjusts to a patient's head, resembling eyeglasses. It features two independent inclinometers, one in the sagittal and one in the frontal plane, and a third in the horizontal plane, indicating head rotation. The device is easy to use, requires minimal palpation, and is affordable compared to more advanced motion analysis systems.
Assessment of impact of neck pain on quality of life | At baseline and after 1 month
  The Neck Bournemouth Questionnaire (NBQ) is a tool measuring neck pain's impact on daily activities and emotional well-being. It covers seven areas and scores 0 to 70, with higher scores indicating greater disability. The NBQ is sensitive and validated in English, French, Dutch, and Arabic.

CONTACTS AND LOCATIONS:
Locations (1):
- outpatient clinic of faculty of physical therapy Benha National university, Banhā, Egypt

IPD SHARING:
Plan to Share IPD: No